CLINICAL TRIAL: NCT04462341
Title: Efficacy of an Oral Hygiene Regimen on Implant Supported, Removable Complete Denture: Effect on Gingival Tissue and Prosthesis: A Proof of Concept Study
Brief Title: Efficacy of an Oral Hygiene Implant Protocol
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Water Pik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 29DRIOH2019
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2020-07

CONDITIONS: Peri-implant Mucositis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Manual brushing only (Active Comparator): Participants brushed with a manual toothbrush and fluoridated toothpaste twice a day for 6 weeks
  Interventions: Device: Manual Toothbrush
- Manual brushing + water flossing (Experimental): Participants brush twice a day and water flossed once a day for 6 weeks.
  Interventions: Device: Water Flosser; Device: Manual Toothbrush

INTERVENTIONS:
Device: Water Flosser — Device that uses water under pressure to clean around teeth and under the gums
  Arms: Manual brushing + water flossing
Device: Manual Toothbrush — Plastic handle with nylon bristles to clean teeth

SUMMARY:
This study is designed to evaluate the effectiveness of cleaning around implants that hold a full denture in the mouth. Different oral hygiene protocols will be compared. Areas to measure are gum tissue color and consistency, bleeding and cleanliness. A questionnaire will be provided at the end of the study. This is a proof of concept study.

DETAILED DESCRIPTION:
The aim of this proof of concept study is to evaluate the effect of an oral hygiene regimen of manual brushing and water flossing on implant retained removable complete dentures. This is a randomized, two arm clinical trial that will compare the traditional oral hygiene regimen to the experimental regimen. Data will be evaluated at baseline, 3 weeks and 6 weeks. Photographs of the tissue and denture will be taken.

ELIGIBILITY:
Inclusion Criteria:

* have a maxillary and/or mandibular implant supported, removable complete denture that is supported by at least 2 implants in good, serviceable condition
* Good general health, with no diseases which could impact periodontal health
* able to read and understand English
* willing to return for all appointments
* at least 30% BOP
* probing depths less or equal to 5mm

Exclusion Criteria:

* subjects who are currently pregnant
* mobility of implant
* subjects who have diabetes
* subjects who smoke
* subjects with any serious medical condition which the investigator feels may impact participation in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing | 6 weeks
  Binary

SECONDARY OUTCOMES:
Probing depth | 6 weeks
  mm

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Kugel, DDS, Study Chair — Tufts School of Dental Medicine
Locations (1):
- Tufts School of Dental Medicine, Boston, Massachusetts, United States